CLINICAL TRIAL: NCT06372522
Title: Continuous Versus Intermittent Oxytocin Infusion for Induction of Labor in Multiparous Pregnant Women
Brief Title: Oxytocin in Multiparous Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Hiba Abu Rass MD, Resident in OB-GYN, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMB-0517-23
Record Dates: First submitted 2024-02-28; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous oxytocin infusion (Experimental): continuous oxytocin infusion - women will continue to receive a continuous oxytocin infusion from start of labor augmentation until delivery.
  Interventions: Drug: Pitocin Injectable Product
- intermittent oxytocin infusion (Active Comparator): intermittent oxytocin infusion - oxytocin transfusion will be discontinued after 8 hours if the woman does not go into active labor, or does not deliver in that period of time.
  The second course of oxytocin will be renewed after 6 hours if the woman hasn't progressed into labor or hasn't given birth yet.
  Interventions: Drug: Pitocin Injectable Product

INTERVENTIONS:
Drug: Pitocin Injectable Product — The primary dose of oxytocin is 1.0 mU/min, with an incremental increase by 2.5 mU/min every 30 minutes, until 20.0 mU/min, tittered to a target of 3-5 contractions in a 10-minute period, or active labor (dilatation > 6 cm).
  Other Names: Synthetic Oxytocin

SUMMARY:
This is a randomized controlled trial investigating whether continuous oxytocin infusion in multiparous women shortens time to delivery, without altering maternal or neonatal outcomes, in augmented deliveries, compared to intermittent infusion.

DETAILED DESCRIPTION:
Induction of labor (IOL) is defined as an artificial initiation of uterine contractions before the spontaneous onset of labor. It is indicated when maternal or fetal risks associated with continuation of pregnancy outweigh the risks associated with early delivery. Augmentation of labor refers to the stimulation of spontaneous but inadequate contractions. In high-income countries, up to 25% of all deliveries at term involve IOL.

Bishop score is a scoring system which measures changes in the cervix. It is based on several characteristics such as cervical effacement, dilatation, consistency, position and fetus head station. A Bishop score < 6 is often referred to as an unripe cervix (unfavorable), whereas ≥ 6 is referred to as a rip cervix (favorable).

Oxytocin is a commonly used drug for IOL, especially in a favorable cervix. It is a mammalian neuro-hypophyseal hormone and is used to generate regular coordinated contractions originating from the fundus towards the cervix. It is administered intravenously (IV) as an increasing infusion, titrated to the strength and frequency of uterine contractions.

There is voluminous experience with oxytocin, and it is considered as a safe drug. Although, there are several case reports reporting rare serious side effects such as: iatrogenic hyponatremia, grand mal seizure and coma, and maternal death. In a prospective observational study of 287 women at term, demonstrated that hyponatremia was correlated significantly with fluid infusion during labor, and not to oxytocin administration.

There is conflicting evidence whether oxytocin infusion should be continued during the active phase of labor or not. Prolonged administration of oxytocin may increase the risk of tachysystole and uterine rupture, which may result in fetal non-reassuring heart rate and caesarian deliveries. Conversely, discontinuing oxytocin infusion after a few hours may have an effect on time to delivery interval, duration of rupture of membrane (ROM) and chorioamnionitis.

one study had shown in an in vitro study that continuous exposure of human myometrial cells to oxytocin led to a loss of responsiveness to oxytocin. Another study, examined myometrial cell cultures from women undergoing cesarean delivery (emergent and elective). They showed that pretreatment of the cells with oxytocin resulted in a decrease in the percentage of myometrial cells that responded to subsequent oxytocin exposure. They found that preliminary exposure of 4.2 hours to oxytocin yielded half-inactivation to the second exposure.

the investigators have previously investigated whether oxytocin infusion duration increases 24-hour delivery rates and affects time to delivery length and patient's experience in nulliparous women. The investigators' results showed that continuous infusion of oxytocin for labor induction in nulliparous women with a favorable cervix may be superior over intermittent oxytocin infusion, since it shortens time-to delivery, decreases chorioamnionitis rate and improves maternal satisfaction, without affecting adverse maternal or neonatal outcomes.

In this study, the investigators' aim is to investigate whether continuous administration of oxytocin is superior to intermittent administration also in multiparous women, in terms of time to delivery and the percentage of women delivering within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* multiparous women (women who have given birth one or more times in the past) with a singleton pregnancy that are admitted for induction of labor.
* Women at gestational age of 370/7 or more.
* Vertex presentation.

Exclusion Criteria:

* Age 18 and under.
* High order gestation.
* Women with contraindication for vaginal delivery.
* Previous cesarean delivery.
* Active labor.
* Documented fetal anomalies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The rate of women delivering within 24 hours. | During admission for delivery (assessed up to 5 days since admission to delivery room)
  number of women (among those who received continues Oxytocin) who manage to deliver within 24 hours from the beginning of the induction.

SECONDARY OUTCOMES:
Length of latent and active phases of labor. | During admission for delivery
  Time interval from admission to delivery room to delivery of fetus
The rate of instrumental and caesarean deliveries. | During admission for delivery
  Cesarean section and operative vaginal delivery including vacuum assisted vaginal delivery
chorioamnionitis | During admission for delivery
  Chorioamnionitis diagnosed at discretion of primary provider during the second stage of labor
obstetric anal sphincter injuries (OASIS) | During admission for delivery
  3rd or 4th degree perineal lacerations
hyponatremia | During admission for delivery
  blood sodium lower than 135 while oxytocin admission
post-partum hemorrhage (PPH) | During admission for delivery
  Estimated blood loss >500 mL for vaginal delivery and >1000 mL for cesarean delivery
neonatal outcome - 1 and 5-minute Apgar score | 1 and 5 minutes after delivery
  apgar score measured at 1 and 5 minutes after delivery
umbilical artery pH | During admission for delivery
  blood withdrawn from umbilical artery after delivery
NICU admission | During admission for delivery
  neonatal admission to ICU unit
Women's satisfaction. | up to 5 days after delivery
  questionnaire - satisfaction scale, with number 1 as the worst score and number 5 as the highest/best score

IPD SHARING:
Plan to Share IPD: No